CLINICAL TRIAL: NCT02500108
Title: Domperidone Use in Parkinson's Disease and Risk of Sudden Cardiac Death
Brief Title: Domperidone and Risk of Sudden Cardiac Death
Status: Completed | Type: Observational
Sponsor: Canadian Network for Observational Drug Effect Studies, CNODES (Other)
Collaborators: Drug Safety and Effectiveness Network, Canada (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Other Study IDs: Q13-02
Record Dates: First submitted 2015-07-14; First posted 2015-07-16 (Estimated); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Parkinson's Disease
Keywords: Domperidone; Ventricular Tachyarrhythmia; Sudden cardiac death; Pharmacotherapy; Adverse events
MeSH Terms: conditions — Parkinson Disease; Tachycardia, Ventricular; Death, Sudden, Cardiac | interventions — Domperidone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Treated with domperidone: Patients who received a new prescription for domperidone (ATC A03FA03) in the year prior to the index date.
  Interventions: Drug: Domperidone
- Unexposed (reference) group: Patients with no prescription for domperidone in the year prior to the index date.

INTERVENTIONS:
Drug: Domperidone — Current exposure to domperidone will be defined as a prescription dispensed within 30 days before the index date.
  Recent exposure to domperidone will be defined as a prescription dispensed between 31 and 90 days before the index date (without a dispensing during the 30 days period preceding index date).
  Past exposure to domperidone will be defined as a prescription dispensed between 91 and 365 days before the index date (without prescription in the 90 days period prior index date).
  Groups: Treated with domperidone

SUMMARY:
The purpose of this study is to assess the risk of serious cardiac events, specifically ventricular tachyarrhythmia and sudden cardiac death (VT/SCD), associated with the use of domperidone in a population of patients with Parkinson's disease. The hypothesis for this study is that the risk of VT/SCD will be higher among domperidone users, especially at a higher dose.

The investigators will conduct a retrospective population-based cohort study using health care databases in eight jurisdictions in Canada and the UK. The study cohort will be defined by the initiation of a new antiparkinsonian drug or a new diagnosis of Parkinson's disease. The results from the separate sites will be combined by meta-analysis to provide an overall assessment of the risk of VT/SCD in users of domperidone.

DETAILED DESCRIPTION:
The purpose of this study is to assess the risk of serious cardiac events associated with the use of domperidone in a cohort of patients with Parkinson's disease. More specifically, the study objective is to assess the risk of ventricular tachyarrhythmia and sudden cardiac death associated with the use of domperidone compared to no use in patients with Parkinson's disease. In addition, the investigators would also like to determine whether the risk of ventricular arrhythmia and sudden cardiac death increases with the dose of domperidone in patients with Parkinson's disease.

The investigators will use a common-protocol approach to conduct retrospective cohort studies using health care data from eight jurisdictions (the Canadian provinces of Alberta, British Columbia, Manitoba, Nova Scotia, Ontario, Quebec, and Saskatchewan, as well as the United Kingdom (UK) Clinical Practice Research Datalink [CPRD]). The Canadian databases contain population-level data on physician billing, diagnoses and procedures from hospital discharge abstracts, vital statistics, and dispensations for prescription drugs. The CPRD is a clinical database that is representative of the UK population and contains the records for patients seen at over 680 general practitioner practices in the UK; these data will be linked to the Hospital Episode Statistics (HES) database, which contains in-hospital diagnosis and procedure data.

Study Population

In each jurisdiction, the investigators will assemble a study cohort that includes all patients with a new diagnosis of Parkinson's disease or a first-ever prescription of an antiparkinsonian drug between January 1, 1990 (or 1 year after site-specific data is available, whichever is later) and June 30, 2012. Patients will be followed from the date of study cohort entry until the occurrence of either study endpoint (defined below) or censoring due to death, departure from the database, loss of continuous health plan or drug plan enrolment, entry into a long-term care facility, or the end of the study period (or the last date of data availability at that site), whichever occurs first. Data from Alberta, Ontario, and Nova Scotia will be restricted to patients aged 66 years and older as prescription data are not available for younger patients.

Case-control selection

The cohort defined above will be analyzed using a nested case-control approach, where cases are defined as a first diagnosis of ventricular tachyarrhythmia (VT) or sudden cardiac death (SCD) any time after cohort entry. For each case, up to 30 controls will be randomly selected among the cohort members in the risk sets defined by the case, after matching on age, sex, date of cohort entry (±1 year), and duration of follow-up. Matching on duration of follow-up (i.e., our best estimate of duration of the disease) will serve as a proxy to control for the potential for confounding by progression and severity of Parkinson's disease.

Exposure Assessment

The clinically relevant exposure period considered for data analysis will be the year preceding the index date, and exposure to domperidone will be classified according to prescriptions dispensed during this time period. For all cases and their matched controls, the investigators will identify all prescriptions for domperidone from the computerized medical records during the year prior to the index date. Current exposure to domperidone will be defined as a prescription dispensed within 30 days before the index date (35 days for Saskatchewan). Recent use, past use, and no use will also be explored as mutually exclusive exposure categories. Recent use will be defined as a prescription dispensed between 31 and 90 days before the index date, and past use as a prescription dispensed between 91 and 365 days before the index date. No use will be defined as no prescription of domperidone in the year preceding the index date and will be the reference category.

Statistical analyses

Conditional logistic regression will be used to estimate the odds ratios and corresponding 95% confidence intervals (CIs) of the association between domperidone use and the risk of VT/SCD. In secondary analyses, VT/SCD will be analyzed according to duration of domperidone use (<=30 days, >30 days), and to the daily dose of domperidone (<=30 mg per day, >30 mg per day). In addition, several sensitivity analyses will be conducted, all defined a priori, to assess the robustness of the results. Finally, all site-specific estimates will be meta-analyzed using fixed and random effects models. The amount of between-site heterogeneity will be estimated using the I square statistic.

ELIGIBILITY:
Inclusion Criteria:

Patients with a diagnosis of Parkinson's disease or a prescription for an antiparkinsonian drug, with at least 365 days of information in the database prior to cohort entry.

Exclusion Criteria:

* Age < 50 on the cohort entry date; or age < 66 in databases with seniors only
* Missing gender
* Less than 1 year of provincial Medicare enrollment and equivalent enrollment in the CPRD preceding cohort entry
* Patients in a long term care facility
* Diagnosis of PD or dispensing (prescription in CPRD) of an antiparkinsonian drug in the year preceding cohort entry
* Patients with a prescription for an antiparkinsonian drug without a diagnosis of Parkinson's disease but with another indication such as atypical Parkinsonism or secondary Parkinsonism, restless legs syndrome, hyperprolactinemia, or acromegaly in the year before cohort entry
* All patients with a prescription for domperidone in the year before cohort entry
* All patients with a history of ventricular tachyarrhythmia, aborted cardiac arrest, implantation of a cardiac defibrillator, cancer other than non-melanoma skin cancer
* Cohort entry date same as cohort exit date (no follow-up)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of all subjects with a diagnosis of Parkinson's disease or a prescription for an antiparkinsonian drug who were registered for provincial medical services coverage or registered in a clinical practice (CPRD) at any time between January 1, 1990 (or 1 year after site-specific data is available, whichever is later) and June 30, 2012.
Sampling Method: Probability Sample
Enrollment: 214962 (Actual)
Dates: Start 2013-05; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Ventricular tachyarrhythmia (VT) or sudden cardiac death (SCD) | Patients will be followed from the date of study cohort entry until the occurrence of VT or SCD, censoring, or for up to 16 years.
  VT/SCD will be defined as patients with one of the following diagnostic codes:
  VT: ICD-9 codes 427.1, 427.4; ICD-10 codes I47.0, I47.2, I49.0. SCD/ cardiac arrest: ICD-9 codes: V12.53, 427.5, 798.1, 798.2, 798.9; ICD-10 codes: Z86.74, I46.0, I46.1, I46.9, R96.0, R96.1, R98.
  All potential cases will be subjected to a computer algorithm to exclude non-relevant events (such as events due to non-arrhythmic cardiac causes or acute life-threatening non-cardiac causes); all potential cases that are not excluded by the algorithm will be reviewed in each centre to exclude cases that do not meet the inclusion and exclusion criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Christel Renoux, MD, PhD, Principal Investigator — Lady Davis Institute for Medical Research, Jewish General Hospital - McGill University
Locations (1):
- Lady Davis Institute for Medical Research, Jewish General Hospital, Montreal, Quebec, Canada

REFERENCES:
- [Result] Renoux C, Dell'Aniello S, Khairy P, Marras C, Bugden S, Turin TC, Blais L, Tamim H, Evans C, Steele R, Dormuth C, Ernst P; Canadian Network for Observational Drug Effect Studies (CNODES) investigators. Ventricular tachyarrhythmia and sudden cardiac death with domperidone use in Parkinson's disease. Br J Clin Pharmacol. 2016 Aug;82(2):461-72. doi: 10.1111/bcp.12964. Epub 2016 May 19. PMID 27062307
- See also: This organization's website describing general functions, other CNODES projects, and investigator profiles. — http://www.cnodes.ca